CLINICAL TRIAL: NCT04373369
Title: A Phase II Study of Maintenance Vorolanib and Atezolizumab in Patients With Extensive-stage SCLC
Brief Title: Vorolanib + Atezolizumab as Maintenance Therapy for Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Funding/Staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202007036
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: Extensive stage small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — vorolanib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vorolanib + Atezolizumab (Experimental): Consenting and eligible participants who have no evidence of tumor progression after 3 to 4 cycles of standard-of-care induction therapy will receive atezolizumab intravenously (IV) every 3 weeks and vorolanib by mouth daily.
  Interventions: Drug: Vorolanib; Drug: Atezolizumab

INTERVENTIONS:
Drug: Vorolanib — Vorolanib is administered orally at a dose of 200 mg on Days 1 through 21 of each 21-day cycle.
  Other Names: X-82
Drug: Atezolizumab — Atezolizumab is administered intravenously at a dose of 1200 mg on Day 1 of each 21-day cycle.
  Other Names: Tecentriq

SUMMARY:
The purpose of the study is to determine whether adding vorolanib to atezolizumab will improve the length of time that participants are cancer-free after receiving standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive stage small cell lung cancer without prior specific systemic therapy aside from induction with platinum, etoposide, and atezolizumab. Measurable disease is not required for eligibility.
* Receipt of at least 3 cycles (and no more than 4 cycles) of platinum plus etoposide and atezolizumab during the induction phase, without tumor progression as determined by CT scan and brain MRI. Patients should be able to start the study treatment no more than 6 weeks from the last dose of induction chemo/immunotherapy. This period may be extended to 8 weeks in patients requiring brain radiotherapy after completion of induction chemo/immunotherapy for brain metastases.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (≤ 5 x IULN for patients with liver metastases)
  * Creatinine ≤ 1.5 x IULN OR measured or calculated creatinine clearance > 50 mL/min for patients with creatinine levels > 1.5 x IULN
  * Urine protein ≤ 1+ or urine protein to creatinine ratio ≤ 1; if UPC ratio is > 1 on urinalysis, then 24-hour urine collection for protein must be obtained and level must be < 1,000 mg for patient enrollment
  * aPTT and either INR or PT ≤ 1.5 x IULN unless participant is receiving anticoagulant therapy as long as PT or a PTT is within therapeutic range of intended use of anticoagulants.
* Patients receiving therapeutic non-Coumadin anticoagulation are eligible, provided they are on a stable dose (per investigator judgment) of anticoagulant.
* The effects of atezolizumab and vorolanib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 31 weeks after last dose of study treatment. Women must use birth control for at least 31 weeks after last dose of study treatment. Women must not be breastfeeding.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria

* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Currently receiving any other investigational agents.
* Patients with untreated brain metastases are excluded. Patients with clinically evident CNS hemorrhage are excluded. Prophylactic cranial irradiation is not allowed. Patients with brain metastases treated with whole brain radiation therapy, radiosurgery, or surgery are eligible.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorolanib, atezolizumab, or other agents used in the study.
* Use of chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* Systemic glucocorticoids with prednisone dose higher than 10 mg/day or equivalent.
* Arterial or venous thromboembolic event, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to enrollment.
* Uncontrolled or poorly controlled hypertension with systolic blood pressure (BP)> 160 mmHg systolic or diastolic > 100 mmHg for > 3 weeks prior to C1D1), despite standard medical management.
* Gastrointestinal perforation, and/or fistula, or risk factors for perforation within 6 months prior to enrollment.
* Grade 3 or 4 gastrointestinal bleeding within 3 months prior to enrollment.
* History of active autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan.
* Hemoptysis (defined as bright red blood or ≥ ½ teaspoon) within 28 days prior to Cycle 1 Day 1 or with radiographic evidence of intratumor cavitation or radiologically documented evidence of major blood vessel invasion or encasement by cancer.
* Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to Cycle 1 Day 1.
* Undergone major surgery within 28 days prior to Cycle 1 Day 1, or minor surgery/subcutaneous venous access device placement within 7 days prior to Cycle 1 Day 1, or has elective or planned major surgery to be performed during the course of the clinical trial.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis at a level of Child-Pugh B or worse, cirrhosis (any degree) with a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis (defined as ascites from cirrhosis requiring diuretics or paracentesis), fatty liver, and inherited liver disease.
* Active tuberculosis.
* Administration of a live, attenuated influenza vaccine within 4 weeks before Cycle 1 Day 1 or at any time during the study.
* Severe infections within 2 weeks prior to Cycle 1 Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to Cycle 1 Day 1. Note: Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* History of deep venous thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to Cycle 1 Day 1.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to C1D1.
* Active hepatitis B (chronic or acute) defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Note: Patients with past or resolved hepatitis B infection (defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test are eligible.
* Patients known to be HIV positive are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2025-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vorolanib + Atezolizumab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vorolanib + Atezolizumab
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 65 [58 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate of Progression-free Survival (PFS) at 6 Months
Description: * Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study.) In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.)
  * Kaplan-Meier product limit estimator will be used to estimate progression-free survival (PFS) at 6 months, with the inclusion of 90% confidence interval.
Time Frame: 6 months
Measure: Number (90% Confidence Interval); unit: percentage of participants-Kaplan Meier
Arm/Group | Vorolanib + Atezolizumab
Number analyzed (Participants) | 11
percentage of participants-Kaplan Meier | 27.3 [8.9 to 49.8]

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: * Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study.) In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.)
Time Frame: Through completion of follow-up for progression-free survival (median length of follow-up 81 days, full range 25-1526 days)
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Vorolanib + Atezolizumab
Number analyzed (Participants) | 11
months | 2.7 [1.3 to 5.1]

3. Secondary Outcome: Median Overall Survival
Description: Overall survival is defined as the length of time from the start of study treatment that patients diagnosed with the disease are still alive.
Time Frame: Through completion of follow-up (median length of follow-up 446 days, full range 93-1526 days)
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Vorolanib + Atezolizumab
Number analyzed (Participants) | 11
months | 14.6 [5.1 to 16.7]

4. Secondary Outcome: Safety and Tolerability of Treatment Regimen as Measured by the Number of Participants With Adverse Events
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Time Frame: From the start of treatment until 90 days after completion of treatment (median length of follow-up 165 days, full range 93-527 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Vorolanib + Atezolizumab
Number analyzed (Participants) | 11
Participants
  Grade 1-2 anemia | 9
  Grade 3-5 anemia | 1
  Grade 1-2 eosinophilia | 1
  Grade 3-5 leukocytosis | 2
  Grade 1-2 sinus tachycardia | 2
  Grade 1-2 vertigo | 1
  Grade 3-5 adrenal insufficiency | 1
  Grade 1-2 allergic conjunctivitis (discharge from eyes due to allergies) | 1
  Grade 1-2 bilateral eye drainage - intermittent | 1
  Grade 1-2 periorbital edema | 1
  Grade 1-2 teeth sensitivity | 1
  Grade 1-2 abdominal pain | 2
  Grade 1-2 bloating | 1
  Grade 1-2 constipation | 1
  Grade 1-2 diarrhea | 5
  Grade 3-5 diarrhea | 1
  Grade 1-2 dry mouth | 1
  Grade 1-2 nausea | 3
  Grade 3-5 nausea | 1
  Grade 3-5 typhitis | 1
  Grade 1-2 vomiting | 3
  Grade 3-5 vomiting | 1
  Grade 1-2 toothache | 1
  Grade 1-2 edema limbs | 3
  Grade 1-2 non cardiac chest pain | 1
  Grade 3-5 generalized weakness | 1
  Grade 1-2 chills | 1
  Grade 1-2 fatigue | 2
  Grade 3-5 fatigue | 2
  Grade 1-2 fever | 3
  Grade 3-5 gait disturbance | 1
  Grade 1-2 malaise | 2
  Grade 3-5 malaise | 1
  Grade 1-2 allergic reaction (poison sumac) | 1
  Grade 1-2 COVID-19 infection | 1
  Grade 1-2 urinary tract infection | 1
  Grade 3-5 lung infection | 2
  Grade 3-5 sepsis | 1
  Grade 1-2 thrush | 1
  Grade 1-2 sunburn | 1
  Grade 1-2 bruising | 1
  Grade 1-2 neutrophil count decreased | 3
  Grade 3-5 neutrophil count decreased | 1
  Grade 3-5 transaminitis | 1
  Grade 1-2 activated partial thromboplastin time prolonged | 4
  Grade 1-2 alanine aminotransferase increased | 5
  Grade 3-5 alanine aminotransferase increased | 1
  Grade 1-2 alkaline phosphatase | 4
  Grade 1-2 aspartate aminotransferase increased | 3
  Grade 3-5 aspartate aminotransferase increased | 1
  Grade 3-5 blood bilirubin increased | 1
  Grade 1-2 blood lactate dehydrogenase increased | 1
  Grade 1-2 creatinine increased | 1
  Grade 1-2 INR increased | 2
  Grade 1-2 lipase increased | 1
  Grade 1-2 lymphocyte count decreased | 3
  Grade 1-2 platelet count decreased | 5
  Grade 3-4 platelet count decreased | 2
  Grade 1-2 white blood cell decreased | 4
  Grade 1-2 malnutrition | 1
  Grade 1-2 anorexia | 4
  Grade 1-2 hyperglycemia | 3
  Grade 1-2 hypertriglyceridemia | 1
  Grade 1-2 hypoalbuminemia | 2
  Grade 1-2 hypocalcemia | 1
  Grade 3-5 hypocalcemia | 1
  Grade 1-2 hypoglycemia | 1
  Grade 1-2 hypokalemia | 1
  Grade 3-5 hypokalemia | 1
  Grade 1-2 hyponatremia | 4
  Grade 3-5 hyponatremia | 1
  Grade 1-2 groin pain | 1
  Grade 3-5 groin pain | 1
  Grade 1-2 muscle aches | 1
  Grade 1-2 arthralgia | 2
  Grade 3-5 back pain | 1
  Grade 3-5 flank pain | 1
  Grade 1-2 generalized muscle weakness | 1
  Grade 3-5 generalized muscle weakness | 1
  Grade 1-2 dizziness | 2
  Grade 1-2 headache | 3
  Grade 1-2 paresthesia | 1
  Grade 1-2 seizure | 1
  Grade 1-2 insomnia | 1
  Grade 1-2 chronic kidney disease (decreased eGFR) | 3
  Grade 1-2 glucosuria | 1
  Grade 1-2 hematuria | 2
  Grade 1-2 proteinuria | 2
  Grade 1-2 orthopnea | 1
  Grade 3-5 acute hypoxemic respiratory failure | 1
  Grade 1-2 allergic rhinitis | 1
  Grade 1-2 cough | 3
  Grade 1-2 dyspnea | 2
  Grade 3-5 dyspnea | 1
  Grade 1-2 epistaxis | 1
  Grade 3-5 hypoxia | 1
  Grade 1-2 pleural effusion | 1
  Grade 1-2 rhinorrhea | 1
  Grade 1-2 sore throat | 1
  Grade 1-2 rash maculo-papular | 1
  Grade 1-2 alopecia | 1
  Grade 1-2 dry skin | 2
  Grade 1-2 hair color changes | 1
  Grade 1-2 pruritus | 1
  Grade 1-2 hypertension | 2
  Grade 3-5 hypertension | 2
  Grade 1-2 hypotension | 1
  Grade 3-5 hypotension | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 90 days after end of treatment (median 165 days, full range 93-527 days). All-cause mortality was followed up to 3 years after discontinuation of study treatment (median 446 days, full range 93-1526 days).
Arm/Group | Vorolanib + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 8/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorolanib + Atezolizumab (N=11)
Adrenal insufficiency (Endocrine disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Lung infection (Infections and infestations) | 2
Platelet count decreased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorolanib + Atezolizumab (N=11)
Anemia (Blood and lymphatic system disorders) | 10
Eosinophilia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Allergic conjunctivitis (discharge from eyes due to allergies) (Eye disorders) | 1
Bilateral eye drainage - intermitten (Eye disorders) | 1
Periorbital edema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Teeth sensitivity (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Typhilitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema limb (General disorders) | 3
Fatigue (General disorders) | 3
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
Generalized weakness (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Allergic reaction (poison sumac) (Immune system disorders) | 1
COVID-19 infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
INR increased (Investigations) | 2
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 6
Transaminitis (Investigations) | 1
Weight loss decreased (Investigations) | 1
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 5
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Muscle aches (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Chronic kidney disease (decreased eGFR) (Renal and urinary disorders) | 3
Glucosuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hair color changes (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04373369/Prot_SAP_000.pdf